CLINICAL TRIAL: NCT01184248
Title: The Effect of Sound Stimulation on Pure-tone Hearing Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Earlogic Korea, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEK14152010
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Sensorineural Hearing Loss
MeSH Terms: conditions — Hearing Loss, Sensorineural

INTERVENTIONS:
Behavioral: Sound stimulation — Listening to sound stimuli at the lowest audible level.

SUMMARY:
The purpose of this study is to investigate if sound stimulation could improve pure-tone hearing threshold.

In the late 1990s, researchers discovered that acoustic stimuli slow progressive sensorineural hearing loss and exposure to a moderately augmented acoustic environment can delay the loss of auditory function. In addition, prolonged exposure to an augmented acoustic environment could improve age-related auditory changes. These ameliorative effects were shown in several types of mouse strains, as long as the acoustic environment was provided prior to the occurrence of severe hearing loss.

In addition to delaying progressive hearing loss, acoustic stimuli could also protect hearing ability against damage by traumatic noise. In particular, a method called forward sound conditioning (i.e., prior exposure to moderate levels of sound) has been shown to reduce noise-induced hearing impairment in a number of mammalian species, including humans.

Interestingly, recent report has suggested that low-level sound conditioning also reduces free radical-induced damage to hair cells, increases antioxidant enzyme activity, and reduces Cox-2 expression in cochlea, and can enhance cochlear sensitivity. Specifically, increased cochlear sensitivity was observed when distortion product otoacoustic emissions (DPOAEs) and compound action potentials (CAPs) were measured.

In addition to forward sound conditioning, backward sound conditioning (i.e., the use of acoustic stimuli after exposure to a traumatic noise) has been shown to protect hearing ability against acoustic trauma and to prevent the cortical map reorganization induced by traumatic noise.

Based on the results of animal studies, the investigators conducted a human study in 2007 and observed that sound stimulation could improve hearing ability. On average, the pure-tone hearing threshold decreased by 8.91 dB after sound stimulation for 2 weeks. In that study, however, the investigators observed only the hearing threshold changes by sound stimulation.

To verify the previous ameliorative effect of sound stimulation, the investigators included a control period in this study.

ELIGIBILITY:
Inclusion Criteria:

* You are a male or female aged between 18 and 70 years
* You have 25~70 dB HL hearing loss at any frequency above 1.5 kHz
* You are able to use an mp3 player
* You are able to read English

Exclusion Criteria:

* Under the medications that could cause hearing loss (such as gentamicin, aspirin, ibuprofen, or acetaminophen)
* Chronic disease that could affect hearing (such as diabetes or high blood pressure)
* Temporal hearing loss
* Hearing loss more than 75 dB HL at any frequency
* Ear infections, chronic middle ear disease or any abnormality of the ear canal or ear drum
* Hearing aid user
* Pregnant females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Changes of pure-tone hearing thresholds after sound stimulation | 4-6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eunyee Kwak, Ph.D., Principal Investigator — Earlogic Auditory Research Institute
Locations (1):
- Earlogic Corporation, Los Angeles, California, United States

REFERENCES:
- [Background] Canlon B, Borg E, Flock A. Protection against noise trauma by pre-exposure to a low level acoustic stimulus. Hear Res. 1988 Jul 15;34(2):197-200. doi: 10.1016/0378-5955(88)90107-4. PMID 3170362
- [Background] Miyakita T, Hellstrom PA, Frimanson E, Axelsson A. Effect of low level acoustic stimulation on temporary threshold shift in young humans. Hear Res. 1992 Jul;60(2):149-55. doi: 10.1016/0378-5955(92)90017-h. PMID 1639725
- [Background] Harris KC, Bielefeld E, Hu BH, Henderson D. Increased resistance to free radical damage induced by low-level sound conditioning. Hear Res. 2006 Mar;213(1-2):118-29. doi: 10.1016/j.heares.2005.11.012. Epub 2006 Feb 8. PMID 16466871
- [Background] Kujawa SG, Liberman MC. Long-term sound conditioning enhances cochlear sensitivity. J Neurophysiol. 1999 Aug;82(2):863-73. doi: 10.1152/jn.1999.82.2.863. PMID 10444683
- [Background] Niu X, Tahera Y, Canlon B. Protection against acoustic trauma by forward and backward sound conditioning. Audiol Neurootol. 2004 Sep-Oct;9(5):265-73. doi: 10.1159/000080226. Epub 2004 Aug 13. PMID 15316199
- [Background] Norena AJ, Eggermont JJ. Enriched acoustic environment after noise trauma reduces hearing loss and prevents cortical map reorganization. J Neurosci. 2005 Jan 19;25(3):699-705. doi: 10.1523/JNEUROSCI.2226-04.2005. PMID 15659607